CLINICAL TRIAL: NCT02258321
Title: A Phase 1, Open-Label, Crossover Study to Evaluate the Relative Bioavailability of a New Tablet Formulation Versus the Current Capsule Formulation of PPI-668 in Healthy Adult Volunteers
Brief Title: Phase 1 Study of Relative Bioavailability of PPI-668 New Tablet Versus Capsule Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Presidio Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PPI-668-104
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Pharmacokinetic Assessments in Healthy Volunteers
MeSH Terms: interventions — ravidasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PPI-668 tablet followed by capsule (Experimental): On day 1, one 200 mg PPI-668 tablet will be administered. On day 6, two 100 mg PI-668 capsules will be administered.
  Interventions: Drug: PPI-668 tablet; Drug: PPI-668 capsule
- PPI-668 capsule followed by tablet (Experimental): On day 1, two 100 mg PI-668 capsules will be administered. On day 6, one 200 mg PPI-668 tablet will be administered.
  Interventions: Drug: PPI-668 tablet; Drug: PPI-668 capsule

INTERVENTIONS:
Drug: PPI-668 tablet
Drug: PPI-668 capsule

SUMMARY:
This study will compare the blood levels of PPI-668 resulting from two different formulations - the current capsule and a new tablet, T003.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to understand and sign a written informed consent form
* nonsmoker
* body mass index (BMI) of 18.0 to 29.9 kg/m2 (inclusive)
* HIV-1 antibody negative.
* hepatitis B (HBV) surface antigen negative.
* hepatitis C (HCV) antibody negative.

Exclusion Criteria:

* Pregnant or lactating subjects.
* Have any serious or active medical or psychiatric illness which, in the opinion of the Investigator, would interfere with subject treatment, assessment, or compliance with the protocol. This would include renal, cardiac, hematologic, hepatic, pulmonary (including chronic asthma), endocrine (e.g., diabetes), central or peripheral nervous, gastrointestinal (including an ulcer), vascular, metabolic (thyroid disorders, adrenal disease), or immunodeficiency disorders, active infection, or malignancy that is clinically significant or requiring treatment.
* Have participated in an investigational trial involving administration of any investigational compound within 30 days prior to the study dosing.
* Current alcohol or substance abuse judged by the Investigator to potentially interfere with subject compliance.
* Have poor venous access and unable to donate blood.
* Have donated blood within 56 days of study dosing.
* Have donated plasma within 7 days of study dosing.
* Have taken any prescription medications or over-the-counter medications including herbal products within 28 days of commencing study drug dosing with the exception of vitamins and/or acetaminophen and/or ibuprofen and/or contraceptive medications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
PPI-668 area under the curve from time zero to infinity (AUC 0-inf) | days 1-8
PPI-668 maximum observed plasma concentration (Cmax) | Days 1-8
PPI-668 area under the curve from time zero to the last quantifiable concentration (AUC 0-t) | Days 1-8

SECONDARY OUTCOMES:
assessments of adverse events | days 1-8
assessments of composite of clinical laboratory parameters | days 1-8

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Brown, MD, Study Director — Presidio Pharmaceuticals
Locations (1):
- Buffalo Clinical Research Center, Buffalo, New York, United States